CLINICAL TRIAL: NCT02841176
Title: A Pilot Study to Evaluate the Utility of Thermography in Assessing Response to Golimumab Treatment in Psoriatic Arthritis
Brief Title: Thermography in Assessing Treatment Response to Golimumab in Psoriatic Arthritis
Acronym: Go-Thermal
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped due to resourcing issues.
Sponsor: Imperial College Healthcare NHS Trust (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16HH3180
Record Dates: First submitted 2016-06-16; First posted 2016-07-22 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2017-08

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Thermography; golimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): Thermography and Golimumab (solution for subcutaneous injection, 50 or 100 mg, monthly)
  Interventions: Other: Thermography; Biological: Golimumab

INTERVENTIONS:
Other: Thermography — Thermographic imaging of arthritic joints will be performed at baseline and within 5 days after the participant's 2nd and 4th doses of monthly Golimumab
Biological: Golimumab — Participants will start monthly Golimumab after their baseline visit

SUMMARY:
This study will be an open label pilot study to explore the utility of thermography in assessing response to Golimumab treatment in Psoriatic Arthritis (PsA). Ten patients fulfilling the Classification criteria for Psoriatic Arthritis (CASPAR) for Psoriatic Arthritis with active disease and eligible for anti-TNF therapy will be invited to participate in this study. They will be assessed at 4 time points during the study: prior to their first anti-TNF medication (screening and basal visits), and subsequently within 5 days after their 2nd and 4th doses of monthly Golimumab.

DETAILED DESCRIPTION:
Psoriatic Arthritis is a joint problem (arthritis) that often occurs with a skin condition called psoriasis. Psoriasis is a common skin problem that causes red patches on the body, and it is an on-going (chronic) inflammatory condition. About 1 in 20 people with psoriasis will develop arthritis with the skin condition. In most cases, psoriasis comes before the arthritis. The cause of Psoriatic Arthritis is not known.

Psoriatic Arthritis can be treated using different types of drugs to reduce pain and swelling of the joints. New medicines that block an inflammatory protein called tumor necrosis factor (TNF) are being widely used for progressive Psoriatic Arthritis, as is the case of the drug Golimumab.

Thermography is the use of images to study heat distribution in different parts of the body, and allows one to see variations in temperature, for example in detecting joint inflammation.

This is a pilot study to evaluate whether thermography is able to reliably detect joint inflammation in Psoriatic Arthritis, and whether it is able to detect improvement or worsening in inflammation during medical treatment with Golimumab. This involves assessing disease activity using some questionnaires, examining of patient joints, performing blood tests, ultrasound and thermography.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 to 95 years
2. Patients fulfilling the CASPAR criteria for Psoriatic Arthritis with active disease
3. Subjects eligible for anti-TNF therapy (ie. have 3 or more swollen and 3 or more tender joints who have failed treatment with 2 disease modifying drugs) and planning to be treated with Golimumab.
4. Subjects may be on oral steroids (prednisone ≤10 mg/day, or equivalent corticosteroid) with a stable dose for the 4 weeks prior to Week 0.
5. Subjects may be on oral NSAIDs with a stable dose for the 4 weeks prior to Week 0.
6. Subjects must be able to adhere to the study visit schedule.
7. The subjects must be capable of giving informed consent and the consent must be obtained prior to any screening procedures.

Exclusion Criteria:

1. Bacterial infections (such as cellulitis), lower respiratory tract infection (such as pneumonia), active tuberculosis infection, viral infections (such as influenza and herpes), bronchitis, sinusitis, superficial fungal infections, abscess. Less serious infections need not be considered exclusions at the discretion of the investigator.
2. Known HIV, Hepatitis B, or Hepatitis C infection.
3. Known hypersensitivity to Golimumab (active substance or to any of the excipients).
4. Allergic reactions (bronchospasm, hypersensitivity, urticaria).
5. Patients who have undergone surgical procedures, including arthroplasty, within the previous year.
6. Latex sensitivity (The needle cover on the prefilled Golimumab pen is manufactured from dry natural rubber containing latex, and may cause allergic reactions in individuals sensitive to latex).
7. Temperature >38.3°C
8. Gastrointestinal inflammatory disorders
9. Asthma and related symptoms (such as wheezing and bronchial hyperactivity)
10. Malignancy within the past 5 years (such as skin cancer, squamous cell carcinoma and melanocytic naevus)
11. Known recent substance abuse (drug or alcohol).
12. Planning to have surgery for PsA or other significant surgery during the period of the study.
13. Participation in another clinical trial involving receipt of an investigational product in the 30 days preceding enrolment, or planned during the study period
14. Unable to undergo any of the study procedures

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-07; Primary Completion 2017-09-19 (Actual); Study Completion 2017-09-19 (Actual)

PRIMARY OUTCOMES:
Temperature over arthritic joint surface, measured by thermography | From baseline up to 97 days

SECONDARY OUTCOMES:
Psoriatic Arthritis Response Criteria (PsARC) | From baseline up to 97 days
Health Assessment Questionnaire (HAQ-DI) | From baseline up to 97 days
Psoriasis Area and Severity Index (PASI) | From baseline up to 97 days
Dermatology Life Quality Index (DLQI) | From baseline up to 97 days
Visual Analog Scale (VAS) assessment of global health | From baseline up to 97 days

CONTACTS AND LOCATIONS:
Overall Officials: Becky Ward, Study Director — Imperial College Healthcare NHS Trust
Locations (1):
- NIHR/Wellcome Trust Imperial Clinical Research Facility, Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available within 1 year of the end of the study